CLINICAL TRIAL: NCT06478017
Title: Belatacept With Delayed Tacrolimus Withdrawal Versus Standard-of-Care Tacrolimus in Heart Transplant Recipients (RTB-013)
Brief Title: Belatacept in Heart Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT RTB-013
Record Dates: First submitted 2024-06-07; First posted 2024-06-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Transplant
Keywords: Heart transplant; Transplantation; Standard of care; Belatacept; Tacrolimus
MeSH Terms: interventions — Abatacept; Tacrolimus; Mycophenolic Acid; Sodium; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belatacept + Tacrolimus withdrawal (Experimental): 1. Maintenance Immunosuppression: NULOJIX (belatacept)
  2. Maintenance Immunosuppression: CellCept (mycophenolate mofetil- MMF), or Myfortic (mycophenolate sodium)
  3. Calcineurin Inhibitors (CNI) Taper: Prograf® (tacrolimus), or tacrolimus generic
  4. Corticosteroid: Prednisone (no less than 5mg per day continued throughout the study period)
  Interventions: Drug: Belatacept; Drug: Tacrolimus; Drug: Mycophenolate Mofetil/Sodium; Drug: Prednisone
- Standard-of-Care (Active Comparator): 1. Maintenance Immunosuppression: Prograf (tacrolimus), or tacrolimus generic;
  2. Maintenance Immunosuppression: CellCept (mycophenolate mofetil- MMF), or Myfortic (mycophenolate sodium);
  3. Corticosteroid +/- taper: Prednisone
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil/Sodium; Drug: Prednisone

INTERVENTIONS:
Drug: Belatacept — Patients will receive 10mg/kg on Day 3 post-transplant (72 hours +/- 12 hours post-transplant)
  Day 7 post-transplant (+/- 6 hours)
  Day 16 (End of Week 2 after 1st dose of belatacept) post-transplant (+/- 2 days)
  Day 30 (End of Week 4 after 1st dose of belatacept) post-transplant (+/- 3 days)
  Day 58 (Week 8) post-transplant (+/- 3 days)
  Day 86 (Week 12) post-transplant (+/- 3 days)
  Patients will receive 5mg/kg Every 28 days (+/- 3 days) thereafter
  Other Names: NULOJIX
  Arms: Belatacept + Tacrolimus withdrawal
Drug: Tacrolimus — Prograf (tacrolimus) or tacrolimus generic
  Other Names: Prograf
Drug: Mycophenolate Mofetil/Sodium — CellCept (mycophenolate mofetil- MMF), or Myfortic (mycophenolate sodium)
  Other Names: CellCept; Myfortic
Drug: Prednisone — Prednisone

SUMMARY:
This is a phase 2, prospective, multi-center, open-label clinical trial. Sixty-six (66) primary heart transplant recipients will be randomized (1:2) to receive either standard-of-care, tacrolimus-based immunosuppression, or a belatacept-based regimen with gradual tacrolimus withdrawal over 9-months post-transplant. Both study arms will receive CellCept® (mycophenolate mofetil- MMF) or Myfortic® (mycophenolate sodium). Corticosteroids will be continued throughout the study in the belatacept arm.

The primary objective is to evaluate whether NULOJIX® (belatacept), when implemented with gradual tacrolimus withdrawal over 9 months, is safe with respect to preventing the composite endpoint of acute cellular rejection (ACR) >= International Society of Heart and Lung Transplantation (ISHLT) 2R, hemodynamic compromise rejection in the absence of a biopsy or histological rejection, re-transplantation, and death at 18 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

Study entry

1. Subject must be able to understand the purpose of the study and be willing to participate and provide written consent
2. Recipient of a primary heart transplant (heart transplant only)
3. Epstein-Barr Virus (EBV) seropositive (VCA IgG, EBNA IgG). If EBNA is not available, enrollment may proceed but the result must be available prior to randomization.
4. Agreement to use contraception; according to the Food and Drug Administration (FDA) Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for the duration of the study
5. In the absence of a contraindication, vaccinations must be up to date per the Division of Allergy, Immunology, and Transplantation (DAIT) Vaccination Guidance for Patients in Transplant Trials (niaidtransplantstudies.org)
6. Mechanical support or investigational drug trials where the intervention ends at the time of transplantation are permitted.

Randomization

1. Recipient of a primary heart transplant
2. No desensitization therapy prior to transplant
3. Negative crossmatch actual or virtual, on the most recent sera as determined by the participating study center
4. Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) prior to randomization
5. Agreement to use contraception; according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for the duration of the study. Those who choose oral contraception must agree to use a second form of contraception after administration of study drug for a period of 1 year after the last dose of study drug
6. Pre-transplant eGFR (CKD-epi) >30ml/min/1.73m^2. If eGFR <30ml/min/1.73m^2 at the time of randomization, participation is permitted if the study physician determines that renal recovery is expected. Participants who are on dialysis at randomization or are expected to require dialysis at or after randomization will not be permitted to participate.

Exclusion Criteria:

Study entry

1. Candidate for multiple solid organ or tissue transplants
2. Prior history of any organ, tissue, or cellular transplant
3. Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow up period
4. History of severe allergic and/or anaphylactic reactions to humanized or murine monoclonal antibodies
5. Known hypersensitivity to NULOIX (belatacept) or ORENCIA (Abatacept)
6. Previous treatment with NULOIX (belatacept) or ORENCIA (Abatacept)
7. Epstein Barr Virus (EBV) seronegative or indeterminant
8. Human Immunodeficiency Virus (HIV) positive
9. Hepatitis B surface antigen positive
10. Hepatitis B core antibody positive
11. Hepatitis C virus antibody (HCV Ab+) and hepatitis C virus (HCV) Polymerase Chain Reaction (PCR) positive patients
12. Patients with active Tuberculosis (TB) in the past 2 years, whether or not it was adequately treated; patients with documented treatment of active TB greater than 2 years ago will be allowed to participate if there is documentation of adequate treatment according to locally accepted clinical practice
13. Subjects must be tested for latent TB infection (LTBI) within a year prior to transplant. Testing should be conducted using either a PPD or Interferon-gamma release assay (i.e., QuantiFERON-TB, T-SPOT.TB). Patients with a positive test for latent TB infection (LTBI) must have completed appropriate therapy for LTBI (https://www.cdc.gov/tb/topic/treatment/ltbi.htm). A subject is considered eligible only if they have a negative test for LTBI within one year prior to transplant OR if they have completed appropriate LTBI therapy within one year prior to transplant
14. Positive serology for T. cruzi or known/suspected history of Chagas disease
15. Participants currently or formerly residing in regions of the US that are highly endemic for coccidiomycosis will undergo serological testing, as per the site's standard of care. Participants with positive serology who have previously been fully treated, will be permitted to participate pending full treatment, and then require prophylaxis as further outlined in Section 7 for the duration of the study. Participants with negative serology who reside in regions where coccidiomycosis is endemic are eligible for enrollment only if they receive prophylaxis for the duration of the study. Endemic regions are determined by site based on local standard of care
16. Findings on pre-transplant or pre-randomization chest x-ray or CT scan suggestive of fungal infection where an alternative etiology is not identified. Participants with a history of positive serologies for histoplasmosis or blastomycosis, performed for clinical indications will be permitted to participate if they have a normal chest x-ray or CT scan but require prophylaxis
17. Known active current viral, fungal, mycobacterial or other infections (including, but not limited to atypical mycobacterial disease and herpes zoster), not including drive line infections
18. Current white blood cell (WBC) count <3.0 or an absolute neutrophil count (ANC) of less than 1500 cells/mm^3 or recurrent leukopenia that is likely to necessitate immunosuppression reduction after transplant, as determined by the site PI
19. History of active inflammatory bowel disease, chronic diarrhea, or malabsorption
20. History of malignancy, per discretion of oncology consult and study oversight team, will be permitted to participate
21. History of AL amyloidosis
22. Patients who are administered or intended to be administered induction therapy (cytolytic agents such as anti-thymocyte globulin or anti-IL2R therapies such as basiliximab) in the immediate peri-transplant period
23. Patients who i) have undergone desensitization, ii) are undergoing or are planned to undergo desensitization, or iii) are intended to receive therapeutic interventions that are used for the purpose of desensitization prior to transplant
24. Pretransplant Calculated Panel Reactive Antibody (cPRA) > 50% as defined by local site practices
25. The use of immunosuppressive biologics within 1 month prior to transplant is not permitted. Non-immunosuppressive biologics such as proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors must be stopped at the time of transplant
26. Patients for whom there is an intent to administer biologics other than those indicated by protocol during the study period
27. The intended use of high dose (>= 2g/kg) intravenous immunoglobulin before or at the time of transplant or before study drug administration
28. A personal history of severe hypogammaglobulinemia (<300mg/dL)
29. Intent to give the patient a live vaccine within 30 days prior to randomization
30. Use or intended use of other investigational drugs after transplant
31. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the potential participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Randomization

1. Recipient of multiple solid organ or tissue transplants
2. Prior history of any organ, tissue, or cellular transplant
3. Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow up period
4. History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies
5. Known hypersensitivity to Belatacept (NULOJIX) or Abatacept (ORENCIA)
6. Previous treatment with Belatacept (NULOJIX) or Abatacept (ORENCIA)
7. Epstein Barr Virus (EBV) seronegative or indeterminant (recipient must be seropositive for VCA IgG and EBNA IgG)
8. HIV positive patient
9. Hepatitis B surface antigen positive patient
10. Hepatitis B core antibody positive patient
11. Hepatitis B negative transplant recipient that received a transplant from a Hepatitis B core antibody positive donor
12. Hepatitis C virus antibody (HCV Ab+) and HCV PCR positive patients
13. Recipient of allograft from a hepatitis C virus nucleic acid test (NAT) positive donor
14. Patients with a previous history of active Tuberculosis (TB) in the past 2 years, whether or not it was adequately treated; patients with documented treatment of active TB greater than 2 years ago will be allowed to participate if there is documentation of adequate treatment according to locally accepted clinical practice
15. Subjects must be tested for latent TB infection (LTBI) within a year prior to transplant. Testing should be conducted using either a PPD or Interferon-gamma release assay (i.e., QuantiFERON-TB, T-SPOT.TB). Patients with a positive test for latent TB infection (LTBI) must complete appropriate therapy for LTBI (https://www.cdc.gov/tb/topic/treatment/ltbi.htm). A subject is considered eligible only if they have a negative test for LTBI within one year prior to transplant OR if they have completed appropriate LTBI therapy within one year prior to transplant
16. Positive serology for T. cruzi or known/suspected history of Chagas disease
17. Participants currently or formerly residing in regions of the US that are highly endemic for coccidiomycosis will undergo serological testing, as per the site's standard of care. Participants with positive serology who have previously been fully treated, will be permitted to participate but require prophylaxis as further outlined in Section 7 of the protocol for the duration of the study. Participants with negative serology who reside in regions where coccidiomycosis is endemic are eligible for enrollment only if they receive prophylaxis for the duration of the study. Endemic regions are determined by site based on local standard of care
18. Findings on pre-transplant or pre-randomization chest x-ray or CT scan suggestive of fungal infection where an alternative etiology is not identified. Participants with a history of positive serologies for histoplasmosis or blastomycosis, performed for clinical indications, will be permitted to participate if they have a normal chest x-ray or CT scan but require prophylaxis as further outlined in Section 7 of the protocol
19. Known active current viral, fungal, mycobacterial or other infections (including, but not limited to atypical mycobacterial disease and herpes zoster), not including drive line infections
20. Current white blood cell (WBC) count <3.0 or an absolute neutrophil count (ANC) of less than 1500 cells/mm^3 or recurrent leukopenia that is likely to necessitate immunosuppression reduction after transplant, as determined by the site PI
21. CMV high risk mismatch (D+/R-)
22. History of active inflammatory bowel disease, chronic diarrhea, or malabsorption
23. History of malignancy, per discretion of oncology consult and study oversight team, will be permitted to participate
24. History of AL amyloidosis
25. Patients who are administered or intended to be administered induction therapy (cytolytic agents such as anti-thymocyte globulin or anti-IL2R therapies such as basiliximab) in the immediate peri-transplant period
26. Patients who have undergone desensitization or received therapeutic interventions that are used for the purpose of desensitization prior to transplant
27. cPRA > 50% at the time of transplant or any donor specific antibodies before or at the time of transplant as determined by local site practices
28. Patients who have been treated with immunosuppressive biologics within 1 month prior to transplant (non-immunosuppressive biologics must have been stopped at the time of transplant)
29. Patients for whom there is an intent to administer biologics other than those indicated by protocol during the study period
30. Patients who are administered or intended to be administered high dose (>=2g/kg) intravenous immunoglobulin in the immediate post-transplant period
31. A personal history of severe hypogammaglobulinemia (<300mg/dL)
32. Receipt of a live vaccine within 30 days prior to randomization
33. Intent to use any other investigational drugs after transplantation
34. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who experience acute cellular rejection (ACR) >ISHLT 2R (local or core read), hemodynamic compromise (HDC) rejection in the absence of a biopsy or histological rejection, re-transplantation, or death as a composite endpoint. | From randomization to 18 months post-transplantation

SECONDARY OUTCOMES:
Slope of estimated glomerular filtration rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) equation | From baseline to 18 months post-transplantation, assessed at Baseline, Randomization, Month 1, 6 and 18
Proportion of subjects with eGFR <60mL/min/1.73m^2 measured by CKD-EPI | From randomization to 18 months post-transplantation
Proportion of subjects with eGFR<45mL/min/1.73m^2 measured by CKD-EPI | From randomization to 18 months post-transplantation
Mean change in albumin/creatinine ratio in urine | From baseline to 18 months post-transplantation
Change in Chronic Kidney Disease (CKD) stage measured using the mean difference on a continuous measurement scale | From Baseline to 18 months post-transplantation, assessed at Baseline, Month 1, 12 and 18
  Chronic Kidney Disease scale:
  Stage 1: Glomerular Filtration Rate (GFR) >90mL/min Stage 2: GFR = 60-89mL/min Stage 3A: GFR=45-59mL/min Stage 3B: GFR=30-44mL/min Stage 4: GFR=15-29mL/min Stage 5: GFR<15mL/min
Proportion of subjects with CKD stage 4 or 5 | From randomization to 18 months, assessed at Month 12 and 18
Mean difference in eGFR between the two arms | 12 months and 18 months
Proportion of subjects who are free from any detection of de novo donor-specific antibodies (dnDSA) | From randomization to 18 months post-transplantation
Number of de novo donor specific antibodies per patient | From randomization to 18 months post-transplantation
Proportion of subjects who are free from ACR greater than or equal to 2R | From randomization to 18 months post-transplantation
Proportion of subjects who are free from ACR 3R | From randomization to 18 months post-transplantation
Proportion of subjects who are free from any treated rejection | From randomization to 18 months post-transplantation
Proportion of subjects who are free from antibody mediated rejection (AMR) (AMR > ISHLT AMR 1) | From randomization to 18 months post-transplantation
Proportion of subjects who are free from hemodynamic compromise rejection in the absence of a biopsy or histological rejection | From randomization to 18 months post-transplantation
Proportion of subjects who are free from mixed rejection (ACR > ISHLT 2R ACR and AMR > ISHLT AMR 1) | From randomization to 18 months post-transplantation
Incidence of acute cellular rejection (ACR) >= International Society of Heart and Lung Transplantation (ISHLT) 2R | From randomization to 18 months post-transplantation
Incidence of acute cellular rejection (ACR) >= International Society of Heart and Lung Transplantation (ISHLT) 3R | From randomization to 18 months post-transplantation
Cumulative incidence of serious infections, including CMV viremia and disease, requiring inpatient/intravenous therapy | From randomization to 18 months post-transplantation
Incidence of post-transplant lymphoproliferative disorder (PTLD) | From randomization to 18 months post-transplantation
Incidence of death | From randomization to 18 months post-transplantation
Incidence of re-listing or re-transplantation | From randomization to 18 months post-transplantation
Incidence of malignancies | From randomization to 18 months post-transplantation
Incidence of interruption/discontinuation of study drug | From randomization to 18 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Joren C Madsen, MD, DPhil, Study Chair — Massachusetts General Hospital; Jon A. Kobashigawa, MD, Study Chair — Cedars-Sinai Medical Center; Marlena Habal, MD, Principal Investigator — NYU Langone Health; Christian P. Larsen, MD, DPhil, Study Chair — Emory University
Locations (4):
- United States (4):
  - Cedars Sinai Heart Institute/ Cedars Sinai Medical (Site # 71146), Los Angeles, California
  - Tampa General Hospital (Site # 71150), Tampa, Florida
  - NYU Langone Health (Site # 71177), New York, New York
  - University of Utah Medical Center (Site # 71126), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait